CLINICAL TRIAL: NCT06196216
Title: Referal Features of Incidental Breast Masses in Chest CT
Brief Title: Breast Lesion in CT Chest
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abeer Mohamed Ali, Doctor, Assiut University
Other Study IDs: CT chest in breast cancer
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MSCT — Enhanced CT chest

SUMMARY:
The aims of this study are To evaluate the CT features of incidental breast lesions on chest CT and subsequently suggest useful criteria for referral to a specialized breast unit.

DETAILED DESCRIPTION:
Enhanced chest CT examination reports containing the key word 'breast' well be reviewed retrospectively. Patients who had incidental breast lesion and were referred to a specialized breast unit and then underwent pathological confirmation well be included. Finally, 100 patients well be enrolled. Two radiologists well evaluate lesion characteristics including; size, shape, margins and enhancement. The correlations between the CT features and pathologies well be evaluated and the diagnostic accuracy of CT features in various combinations well be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patients who ex hibited incidental breast lesion(s) on enhanced chest CT and were referred to a specialized breast unit for assessment and then underwent pathological confirmation.

Exclusion Criteria:

* -Patients with known breast dis ease.
* Previous history of breast cancer or breast surgery.
* Patients who had undergone only non-enhanced CT examination.

Ages: 25 Years to 95 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult female
Study Population: adult female patients who underwent enhanced CT chest that incidentally revealed breast lesion(s) then referred to a specialized breast centre and had histopathological diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
detect useful CT criteria of breast lesions subsequently suggest criteria for referral to a specialized breast unit | 3years
  detect useful CT criteria of breast lesions subsequently suggest criteria for referral to a specialized breast unit

CONTACTS AND LOCATIONS:
Overall Officials: Abo-Elhassan Hassib Mohamed, Associate professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Harish MG, Konda SD, MacMahon H, Newstead GM. Breast lesions incidentally detected with CT: what the general radiologist needs to know. Radiographics. 2007 Oct;27 Suppl 1:S37-51. doi: 10.1148/rg.27si075510. PMID 18180233